CLINICAL TRIAL: NCT06968455
Title: The Association of Endocrine Disruptors and Toxic and Essential Chemical Elements With Polycystic Ovary Syndrome
Brief Title: Endocrine Disruptors, Toxic and Essential Chemical Elements and Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: TP20220007
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; endocrine disrupting chemicals; bisphenol A; parabens; triclosan; heavy metals
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Parabens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — • venous blood, first morning urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS study group: PCOS patients aged 20 to 39 years
  Interventions: Other: parabens
- healthy control group: Healthy women aged 20 to 39 years
  Interventions: Other: parabens

INTERVENTIONS:
Other: parabens — endocrine disruptors

SUMMARY:
Studies have shown that endocrine disruptors (EDs) and toxic and essential chemical elements affect women's reproductive health and may play a role in the development of polycystic ovary syndrome (PCOS). There is little research examining the association of EDs and toxic and essential chemical elements with PCOS, and for some chemical compounds there is none. In our study, we will examine the relationship of EDs (bisphenols, parabens, triclosan) and toxic (cadmium-Cd, lead-Pb, mercury-Hg, arsenic-As) and essential chemical elements (selenium-Se, copper-Cu, zinc-Zn, manganum-Mn, molibdenum-Mo) in biological samples (blood, urine) of women with PCOS. Main hypothesis is that the levels of EDs, toxic chemical elements and molibdenum-Mo in the biological samples of PCOS women will be higher, and the levels of essential chemical elements will be lower than in the control group and related to the altered liver and kidney function and to the women's lifestyle and the environment they live in.

DETAILED DESCRIPTION:
Endocrine disruptors are externally introduced chemical substances or mixtures of substances that, through altering hormone functions, cause unwanted effects on the health of an individual or its offspring or (sub)population. They are ubiquitous in the environment in polycarbonate plastic and plastic packaging (bisphenols) or in cosmetic and pharmaceutical products (parabens, triclosan). They enter the body through food and drinking water consumption, through inhaled air and contact with the skin. Studies have shown that EDs, especially bisphenols (e.g., bisphenol A-BPA, bisphenol S-BPS, bisphenol F-BPF), parabens and triclosan, through their impact on steroid receptors and epigenetic modifications, have a negative effect on women's reproductive health. Exposure to toxic and essential chemical elements can trigger the formation of reactive oxygen species, which affects steroidogenesis and metabolic processes.

The heterogeneity of the clinical picture in PCOS suggests that, in addition to genetic factors, environmental factors and lifestyle might also be involved in the etiopatoghenesis of the syndrome. Therefore, EDs are also the subject of research for a possible role in the development of PCOS. Some studies have confirmed elevated levels of BPA in the blood and urine of women with PCOS. The positive correlation of BPS with PCOS has been confirmed in only one study so far. The only study assessing blood levels of parabens in women with PCOS found no association with PCOS. So far, only two studies have examined the association of triclosan with PCOS, with conflicting results. Elevated levels of toxic chemical elements (e.g., Cd, Pb, Hg, As) and reduced levels of essential elements (e.g., Se, Zn) can also play a role in the development of PCOS. There are no studies assessing the role of Mo in PCOS. Since the current data on association of EDs and toxic and essential chemical elements with PCOS is scarce, the information obtained in our research could allow us to give an expert opinion on additional diagnostic tests and future recommendations on how to avoid the negative impact of EDs, toxic and essential chemical elements.

The research will be conducted at the Division of Obstetrics and Gynaecology, University Medical Centre Ljubljana, with the collaboration of the Clinical Research Centre, University Medical Centre Ljubljana, Institute of Clinical Chemistry and Biochemistry, University Medical Centre Ljubljana, and Jožef Stefan Institute. The study will be a prospective case-control study. The required number of samples was estimated based on one of the few published studies, where the presence of BPA was found in 95 % of PCOS women, while in the control group this proportion was 70 %. When analyzing the study power, we considered the standard values for alpha = 0.05 and a power of 80%. With these assumptions, we would need 35 women in each group. Women will be introduced to the study when treated for PCOS (study group) or attending the Division of Obstetrics and Gynaecology, University Medical Centre Ljubljana, for a regular periodic gynecological check-up (control group). After signing the informed consent form, clinical examination and transvaginal ultrasound with the antral follicle count will be performed. Each woman will fill in the questionnaire regarding her health status, fertility, pregnancies, deliveries, region of permanent residence, home and workplace environment, dietary and lifestyle habits, smoking and education. On the day 2 to 5 of regular menstrual cycle or after two or more months after last menstrual period in the case of oligo- or amenorrhea, fasting venous blood sample and first morning urine will be taken at the Institute of Clinical Chemistry and Biochemistry, University Medical Centre Ljubljana, for analysis of the content of bisphenols (BPA, BPS and BPF), parabens, triclosan, chemical elements (toxic - Cd, Pb, Hg and As, and essential - Se, Cu, Zn, Mn, Mo), blood count, liver and kidney function tests, Antimüllerian hormone-AMH, sex hormone binding globuline- SHBG and reproductive hormones (FSH, LH, PRL, TSH, estradiol, progesterone, testosterone, androstenedione, dehydroepiandrosterone sulfate). The analysis of EDs and chemical elements will be carried out at the Jožef Stefan Institute, while other diagnostic tests will be carried out at the Clinical Institute for Clinical Chemistry and Biochemistry, University Medical Centre Ljubljana, where the collection of biological samples will also take place. The protection of personal data will be guaranteed, as each blood sample will be labelled or recorded during the study under a code identical to the code of the questionnaire completed by the patient. The statistical evaluation of the data will be carried out at the University Medical Centre Ljubljana, Jožef Stefan Institute, and the Faculty of Medicine, University of Ljubljana. Appropriate statistical models, e.g., multiple linear regression, will be used to determine the relationship between EDs exposure, PCOS and lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18.5 and 29.9 kg/m2
* fulfilling two of the three Rotterdam diagnostic criteria for the diagnosis of PCOS: oligo- or anovulation, ultrasound-visible morphological picture of PCO (presence of 12 or more follicles of size 2-9 mm in one of the ovaries) and/or clinical/biochemical signs of hyperandrogenism (study group)
* a regular menstrual cycle of 21 to 35 days (control group)

Exclusion Criteria:

* pregnancy
* hormonal treatment in the last 3 months (hormonal contraception, hormone replacement therapy, progestogens)
* hyperprolactinemia
* hypothyroidism, hyperthyroidism
* known premature ovarian failure, primary amenorrhea
* chronic diseases: diabetes, depression, Crohn's disease, celiac disease, cardiovascular diseases, liver and kidney disease, asthma, chronic obstructive pulmonary disease, diseases of the musculoskeletal system, neurological diseases, oncological diseases.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women attending the Division of Ob/Gyn, University Medical Centre Ljubljana, for PCOS treatment or a regular periodic gynecological check-up.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Levels of EDs, toxic and essential chemical elements in biological samples (blood, urine) | 1 month
  blood and urine levels

SECONDARY OUTCOMES:
liver and kidney function | 1 month
  biochemical testa
reproductive hormone blood levels | 1 month
  blood levels

CONTACTS AND LOCATIONS:
Overall Officials: Irma Virant-Klun, PhD, Principal Investigator — Clinical Research Centre, University Medical Centre Ljubljana
Locations (1):
- Division of Ob/Gyn, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Rattan S, Zhou C, Chiang C, Mahalingam S, Brehm E, Flaws JA. Exposure to endocrine disruptors during adulthood: consequences for female fertility. J Endocrinol. 2017 Jun;233(3):R109-R129. doi: 10.1530/JOE-17-0023. Epub 2017 Mar 29. PMID 28356401
- [Background] Yilmaz B, Terekeci H, Sandal S, Kelestimur F. Endocrine disrupting chemicals: exposure, effects on human health, mechanism of action, models for testing and strategies for prevention. Rev Endocr Metab Disord. 2020 Mar;21(1):127-147. doi: 10.1007/s11154-019-09521-z. PMID 31792807
- [Background] Chiang C, Mahalingam S, Flaws JA. Environmental Contaminants Affecting Fertility and Somatic Health. Semin Reprod Med. 2017 May;35(3):241-249. doi: 10.1055/s-0037-1603569. Epub 2017 Jun 28. PMID 28658707
- [Background] Ye J, Zhu W, Liu H, Mao Y, Jin F, Zhang J. Environmental exposure to triclosan and polycystic ovary syndrome: a cross-sectional study in China. BMJ Open. 2018 Oct 17;8(10):e019707. doi: 10.1136/bmjopen-2017-019707. PMID 30337305
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5295269/